CLINICAL TRIAL: NCT04303143
Title: Hypnosis and Direct Autonomic Experience Influence on Chronic Symptoms
Acronym: HDAX1
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Inner Group Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: HypDax1
Record Dates: First submitted 2020-03-07; First posted 2020-03-10 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Restless Legs Syndrome; Multiple Sclerosis; Trauma, Psychological; Chronic Disease; Trauma
Keywords: hypnosis; trauma; chronic disease
MeSH Terms: conditions — Restless Legs Syndrome; Multiple Sclerosis; Psychological Trauma; Chronic Disease; Wounds and Injuries | interventions — Hypnosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Primary: Primary
  Interventions: Behavioral: Self-Hypnosis; Behavioral: Direct Autonomic Experience Control

INTERVENTIONS:
Behavioral: Self-Hypnosis — Self-Hypnosis
Behavioral: Direct Autonomic Experience Control — Direct Autonomic Experience Control. Use of learned mental tool/process to affect outcome measure of SUDS discomfort experience. (eg. Squeeze hand as pre-learned mental anchor to relieve discomfort in lower legs)
  Other Names: DAX Control

SUMMARY:
Study will look at a limited number of participants with various chronic symptoms. Investigating a new and novel form of hypnosis application called "Direct Autonomic Experience (DAX)" which is using combination of visualization, metaphor, post-hypnotic suggestion and anchoring.

Purpose is to confirm that DAX generally appears to impact SUDS value and subjects report observed level of effect on short and longer term measurements.

Most significantly, testing that DAX technique/action is reusable later if the measured SUDS value returns or increases.

DETAILED DESCRIPTION:
Hypnosis and Direct Autonomic Experience Influence on Chronic Symptoms One common characteristic of many chronic conditions is the neurology/ biology/ symptomology may change slightly or signficantly over time. So an initial process/plan that worked well for affecting a SUDS discomfort level, may no longer work or work as well.

DAX is designed to be adaptive such that as matters that affected the initial SUDS conditions may have changed, shifted, grown or otherwise be different.

(Examples are increased lesions with MS). Where initial patterns were created with a certain set of neural condition and pathways. But now days/weeks later, with new pathways created, can a previously installed DAX pattern adjust and shift to accommodate the new neural patterns based on participants willingness and self-instruction, or does it require professional adjustment.

Example participant given strong post-hypnotic suggestions/anchor/etc to squeeze right hand in certain way to bring relief to leg discomfort. Initial testing shows working. Now time has shifted, maybe new pathways or other chronic conditions have changed. Can the DAX processes the participant has been taught handle these changes or does it require a professional to re-apply/boost or incorporate new details to get significant changes to reported SUDS discomfort values.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have a proper medical diagnosis of chronic condition.
* Existing medical treatments are having little to no effect on a discomfort metric to measure
* SUDS to be evaluated could be physical or emotional in nature (e.g. Anxiety level, or Leg Cramping/moving)
* Must be motivated and willing to participate in a study that uses hypnosis, placebo and/or nocebo type mental matters.
* Participant must continue existing medical treatments (as recommended/adjusted by such outside professionals) and continue to see and be monitored by new/existing medical professionals during the term of study.
* Must have technology of computers/internet/support to be able to attend regular video chat/conferences for needed interactions with study.
* Must have schedule availability and flexibility to meet in video chats/conferences as required.
* Must have the computer skills/resources and aptitude to handle video chat/conference and able to have resources/friends/knowledge that can help if technical issues arise to allow conference to occur (can handle restarting a video conference if crashes or network acts up)

Exclusion Criteria:

* Acute and short term discomfort matters not being measured that outside scope of chronic condition.
* Must not be active in any other studies or such studies deemed to not interact with this.
* Does not have a properly diagnosed chronic condition (exception are control subjects)

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Open to anyone over age or 12 (with proper adult/guardian supervision/authorization) with a proper medical chronic condition with one discomfort item (may have many, but only picking one) to be measured and evaluated over term of this study
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
SUDS | 7 days
  Subject Unit of Discomfort Symptom. Each patient will have different types and levels of discomfort. Could be back, legs, whatever. Once identified and a numerical value applied to level of discomfort on scale of 1 to 10. We will track that particular SUDS metric through the study, looking for various factors that enable the measured value to drop to lowest value and to re-correct back to lower value if conditions cause it to rise again.

SECONDARY OUTCOMES:
DAX Control of SUDS Change | 1 day
  Direct Autonomic Experience (DAX) is patients ability to use pre-learned applied conscious and subconscious controls to their specified Subject Unit of Discomfort Symptom (SUDS) Discomfort related to their chronic condition. (self-adjustment). Comparing what patient can do on own, compared to when professional doing same to impact the identified SUDS discomfort item.
Professional Control of SUDS change | 1 day
  Participants ability to use pre-learned applied conscious and subconscious controls to their specified Subject Unit of Discomfort Symptom (SUDS) Discomfort related to their chronic condition with professional assistance (professional-adjustment)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Vendemia, BCH, MNLP, Principal Investigator — Inner Group Inc.

IPD SHARING:
Plan to Share IPD: No